CLINICAL TRIAL: NCT05916040
Title: Total Neoadjuvant Treatment of Rectal Cancer by MRI-guided Radiotherapy: a Prospective Observational Study
Brief Title: Total Neoadjuvant Treatment of Rectal Cancer by MRI-guided Radiotherapy
Acronym: TNTRect
Status: Recruiting | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Mark De Ridder, Principal Investigator, Prof., Universitair Ziekenhuis Brussel
Other Study IDs: TNTRect
Record Dates: First submitted 2023-05-24; First posted 2023-06-23 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Rectal Cancer
Keywords: Radiation therapy; MR-guided radiotherapy; Stereotactic body radiotherapy; Total Neo-adjuvant Treatment
MeSH Terms: conditions — Rectal Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- TNTRect MRI-guided radiotherapy group with simultaneous integrated boost: Interventions include having received MRI-guided therapy with simultaneous integrated boost on the gross tumor volume in patients with rectum cancer.
  Interventions: Device: Radiotherapy with MRIdian with simultaneous integrated boost; Other: Questionnaires before, during and after radiotherapy

INTERVENTIONS:
Device: Radiotherapy with MRIdian with simultaneous integrated boost — radiotherapy during 5 days given in 5 weekdays with simultaneous integrated boost
  Other Names: Radiotherapy with MRIdian (ViewRay Inc.)
Other: Questionnaires before, during and after radiotherapy — Questionnaires consisting of 3 quality of life scales and 1 mental state scale:
  * EORTC QLQ-C30
  * EORTC QLQ-CR29
  * Low Anterior Resection Syndrome Score (LARS) questionnaire
  * Hospital Anxiety and Depression Scale (HADS) questionnaire

SUMMARY:
The TNTRect trial is a prospective observational study that will evaluate the outcome of MR-guided stereotactic body radiotherapy (SBRT) with a simultaneous integrated boost in a hypofractionated treatment of rectum cancer. Patients will be treated in 5 daily fractions of 5 Gy within an overall treatment time (OTT) of 5 days. A simultaneous integrated boost (SIB) till 30Gy will be delivered to the gross tumor volume. Patients will be treated with daily adaptive radiotherapy and online tumor gating on the MRIdian system (ViewRay Inc.). The aim of the study is to improve the complete clinical response rate to offer more patients an organ preserving approach.

The primary endpoint is patient response to the treatment, assessed by endoscopy and MRI, or by medical pathology reports after potential resection was performed. As secondary endpoints local control, disease-free survival, overall survival and the patient's quality of life & hospital anxiety and depression will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced rectal cancer

Exclusion Criteria:

* Patients with unresectable metastatic disease at diagnosis
* Patients with an ECOG performance status > 2
* Patients not deemed fit for radiotherapy, chemotherapy or surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with rectal cancer aged 18 years or older.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2024-11-28 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Response to therapy | up to 25 weeks after start of radiotherapy
  After radiotherapy and chemotherapy are administered, the patient will be evaluated for a potential watchful-waiting approach where, together with the patient, can be opted too not perform a TME (total mesorectal excision). This outcome measure registers if the therapy works.

SECONDARY OUTCOMES:
Quality of life assessment via QLQ-C30 | from the start of radiotherapy until 5 years after treatment
  Quality of life according to EORTC Quality of life Questionnaire QLQ-C30
Colorectal specific quality of life assessment via QLQ-CR29 | from the start of radiotherapy until 5 years after treatment
  Colorectal specific quality of life according to EORTC Quality of life Questionnaire QLQ-CR29
Bowel functioning specific quality of life assessment via LARS score | from the start of radiotherapy until 5 years after treatment
  Bowel functioning quality of life according to Emmertsen and Lauberg's[1] Quality of life Questionnaire LARS.
  [1]: Emmertsen KJ, Laurberg S. Low anterior resection syndrome score: development and validation of a symptom-based scoring system for bowel dysfunction after low anterior resection for rectal cancer. Ann Surg. 2012;255:922-8.
  In that scientific publication, the authors introduced a practical and psychometrically robust instrument for examining bowel function (after surgery in rectal cancer), which reflects impact on quality of life.
Anxiety and depression state via HADS | from the start of radiotherapy until 5 years after treatment
  Hospital Anxiety and Depression Scale (HADS) according to Zigmond and Snaith [2].
  [2]: Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70.
  In that scientific publication, the authors introduced a self-assessment scale to be a reliable instrument for detecting states of depression and anxiety in the setting of an hospital medical outpatient clinic.

CONTACTS AND LOCATIONS:
Overall Officials: Mark De Ridder, MD, Principal Investigator — Department of Radiotherapy, UZ Brussel, Vrije Universiteit Brussel
Locations (1):
- UZ Brussel - Dienst Radiotherapie, Jette, Brussels Capital, Belgium